CLINICAL TRIAL: NCT03082937
Title: An Open Label, Single-Dose, Single Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-A4250 in Healthy Male Subjects
Brief Title: An Open Label, Single-dose, Single Period ADME Study of A4250 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4250-007; 2016-002923-27 (EudraCT Number)
Record Dates: First submitted 2017-02-27; First posted 2017-03-17 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Orphan Cholestatic Liver Diseases; Progressive Familial Intrahepatic Cholestasis; Alagille Syndrome; Primary Biliary Cirrhosis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Alagille Syndrome; Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 mg [14C]-A4250 capsule (Experimental)
  Interventions: Drug: 3 mg [14C]-A4250 capsule

INTERVENTIONS:
Drug: 3 mg [14C]-A4250 capsule — Each subject will receive a single administration of 3 mg [14C]-A4250 capsule for oral administration containing not more than 4.3 MBq (116 μCi), in the fasted state.

SUMMARY:
The primary objectives of the study are to assess the mass balance recovery after a single dose of carbon-14 [14C]-A4250 as a capsule and to provide plasma, urine and faecal samples for metabolite profiling and structural identification in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 30 to 65 years of age
3. Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Must be willing and able to communicate and participate in the whole study
5. Must have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day)
6. Must provide written informed consent
7. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months prior to screening
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who have smoked within the last 12 months. A confirmed positive urine cotinine test at screening or admission
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
10. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
11. Confirmed positive drugs of abuse test result at screening or admission
12. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
13. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <90 mL/min using the Cockcroft-Gault equation
14. History of cardiovascular, renal, hepatic, chronic respiratory or GI disease as judged by the investigator
15. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
16. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
17. Donation or loss of greater than 400 mL of blood within the previous 3 months
18. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
19. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
To assess mass balance recovery of total radioactivity in urine | Between pre-dose (admission to 0 hour) and post dose (ending on morning of discharge (up to day 10 depending on if mass balance cumulative recovery >90% or <1% of dose has been collected))
  Amount excreted (Ae) and Ae as a percentage of the administered dose (% Ae), cumulative recovery (CumAe) and cumulative recovery expressed as a percentage of the dose (Cum%Ae)
To assess mass balance recovery of total radioactivity in faeces | Between pre-dose (admission to 0 hour) and post dose (ending on the morning of discharge (up to day 10 depending on if mass balance cumulative recovery >90% or <1% of dose has been collected))
  Amount excreted (Ae) and Ae as a percentage of the administered dose (% Ae), cumulative recovery (CumAe) and cumulative recovery expressed as a percentage of the dose (Cum%Ae)
Metabolite profiling of A4250 of plasma using liquid-chromatography-radio-detection with subsequent mass spectrometry as appropriate | Between pre-dose and up to 48 hours post dose
  Identification of the chemical structure of each metabolite accounting for greater than 10% of circulating radioactivity in plasma
Metabolite profiling of A4250 of urine using liquid-chromatography-radio-detection with subsequent mass spectrometry as appropriate | Between pre-dose (admission to 0 hour) and post dose (ending on the morning of discharge (up to day 10 depending on if mass balance cumulative recovery >90% or <1% of dose has been collected))
  Identification of the chemical structure of each metabolite accounting for greater than 10% of the dose in urine
Metabolite profiling of A4250 of faeces using liquid-chromatography-radio-detection with subsequent mass spectrometry as appropriate | Between pre-dose (admission to 0 hour) and post dose (ending on the morning of discharge (up to day 10 depending on if mass balance cumulative recovery >90% or <1% of dose has been collected))
  Identification of the chemical structure of each metabolite accounting for greater than 10% of the dose in faeces

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No